CLINICAL TRIAL: NCT04888091
Title: The Effect of Two Different Cervical Mucus Removal Methods on Pregnancy Rates. 180 Cases Will be Randomized Into 3 Groups for Cervical Mucus Intervention. Removal With Cotton Swab, Removal With Cannula and Mucus Left on Cervix.
Brief Title: Comparison of the Effect of Cervical Mucus Cleaning Method Applied Before Embryo Transfer on Pregnancy Rates.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, enis ozkaya, Associate Professor, Specialist in Obstetrics and Gynecology, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90-07.April.2021
Record Dates: First submitted 2021-05-03; First posted 2021-05-17 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Infertility
Keywords: Cervical mucus; Embryo transfer; Pregnancy rate
MeSH Terms: conditions — Infertility | interventions — Cannula

STUDY DESIGN:
Intervention Model Description: It is a parallel model interventional study. The sample size is calculated as 180 patients. Sixty patients will be assigned to each study arm by randomization. It is planned to use random computerized numbers for randomization. İn arm 1, cervical mucus will be removed with a cotton swab before embryo transfer. In arm 2, cervical mucus will be removed with a canula before embryo transfer. In arm 3, cervical mucus will not be removed.
Who Masked: Participant
Masking Description: Participant masking: Embryo transfer is done while the patient is lying in lithotomy position in accordance with gynecological examination. The patient is informed about the preparations before the embryo transfer and then the examination is completed. The patient will not be informed about the method used for removal of the cervical mucus. The patient's lying position also does not allow observation of the material used to remove cervical mucus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cervical mucus removal with cotton swab (Active Comparator): Cervical mucus will be removed with cotton swab before embryo transfer
  Interventions: Procedure: Cotton swab
- Cervical mucus removal with cannula (Active Comparator): Cervical mucus will be removed with cannula before embryo transfer
  Interventions: Procedure: Cannula
- No cervical mucus removal (No Intervention): Cervical mucus will not be removed prior to embryo transfer

INTERVENTIONS:
Procedure: Cotton swab — Removal of the cervical mucus with a cotton swab before embryo transfer.
  Arms: Cervical mucus removal with cotton swab
Procedure: Cannula — Removal of the cervical mucus with a cannula before embryo transfer.
  Arms: Cervical mucus removal with cannula

SUMMARY:
To assess the impact of cervical mucus cleansing before embryo transfer and compare two different instruments for this purpose.

DETAILED DESCRIPTION:
All patients will be informed about the study and those who give written consent will be included in the study.

Women undergoing good quality embryo transfer will be assigned to one of the 3 arms of the study according to the previously determined randomization chart. The first evaluation of the patient will be made on the 12th day after embryo transfer. Pregnancy status will be evaluated with serum βhcg value. If pregnancy is confirmed by serum βhcg value, fetal viability will be evaluated by ultrasound 4 weeks after transfer.

ELIGIBILITY:
Inclusion Criteria:

* 21-40 years old women,
* Women undergoing good quality embryo transfer,
* Women who are eligible for a single or double embryo transfer.

Exclusion Criteria:

* If there is a diagnosis of a uterine anomaly,
* If there is a diagnosis of myoma uteri,
* If there is a diagnosis of rheumatological disease,
* Women to be transferred other than good quality embryo,
* Hİstory of previous pelvic, gynecological operation.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Detecting pregnancy after embryo transfer. | 12 days after embryo transfer/ intervention.
  Confirmation of pregnancy with serum βhcg value at the earliest 12th day after embryo transfer.
Confirmation of fetal cardiac activity in detected pregnancy. | 3-4 weeks after embryo transfer/ intervention.
  Evaluation of fetal cardiac activity on ultrasound.

SECONDARY OUTCOMES:
Success of embryo transfer during intervention. | 5 minutes after embryo transfer.
  In some cases, the embryo is transferred to the endometrial cavity and comes back with the transfer cannula. For this reason, the embryology laboratory checks the transfer cannula after the transfer. If the embryo is still in the embryo transfer cannula, a second attempt is made for embryo transfer. As a secondary outcome, we will evaluate the success in the first attempt for embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Belgin Devranoğlu, Ass. Prof., Principal Investigator — Zeynep Kamil Women and Children's Diseases Training and Research Hospital; Müşerref Banu Yılmaz, Md., Study Director — Zeynep Kamil Women and Children's Diseases Training and Research Hospital
Locations (1):
- Zeynep Kamil Women and Children's Diseases Training and Research Hospital, Istanbul, Turkey (Türkiye)